CLINICAL TRIAL: NCT05634031
Title: Development and Validation of a Non-invasive Algorithm for Diagnosis of Microvascular Angina Among Patients With Ischemia and Non-obstructive Coronary Artery Disease (IMAGING-CMD Study)
Brief Title: Imaging Coronary Microvascular Dysfunction (CMD) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Krishna Patel, Assistant Professor of Medicine (Cardiology) and Population Health Science and Policy, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY-22-00774; IF2779994 (Other Grant/Funding Number: Jubilant DraxImage, Inc.)
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Angina; Non-obstructive Coronary Artery Disease
MeSH Terms: conditions — Angina Pectoris | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with INOCA (Experimental): Patients to undergo coronary angiogram and/or coronary CT angiogram for suspected ischemic symptoms of angina and dyspnea but do not have obstructive epicardial coronary artery disease.
  Interventions: Radiation: PET imaging; Radiation: Coronary CT angiogram; Procedure: Functional Angiography; Procedure: Treadmill exercise stress study

INTERVENTIONS:
Radiation: PET imaging — PET imaging visit, which will take approximately 1-2 hours.
Radiation: Coronary CT angiogram — A coronary CT angiogram if the participant has not had one recently.
Procedure: Functional Angiography — A subset of patients with abnormal results on cardiac PET myocardial perfusion imaging study (estimated number of patients = 12) will be invited to participate in an invasive sub-study wherein they would undergo detailed invasive coronary physiology evaluation.
  Functional Angiography (coronary reactivity test- CRT): is an angiography procedure done in the catheterization laboratory. It evaluates the coronary artery microcirculation and how the blood vessels respond to different medications.
  Other Names: coronary reactivity test; CRT
Procedure: Treadmill exercise stress study — A treadmill exercise stress study

SUMMARY:
Angina is a common clinical symptom of ischemic heart disease, affecting up to 11 million people in the United States alone, and 112 million people globally. Despite this, 4 in 10 patients undergoing elective coronary angiography for angina and ischemia do not have evidence of obstructive coronary artery disease (CAD). This condition of ischemia with no obstructive CAD (INOCA) is associated with high clinical and economic morbidity, as these patients have a higher rate of repeat procedures and hospitalizations, worse quality of life, future adverse cardiovascular events and frequent time missed from work.

The overall objective of this study is to develop and validate a non-invasive algorithm for diagnosis and management of patients with INOCA and suspected microvascular dysfunction centered around cardiac PET MPI. A secondary goal of the study is to assess for improvement in patient symptoms, function and quality of life from PET-guided management of CMD in patients with INOCA.

This study will take place at Mount Sinai Morningside in the PET and CTunit on the 3rd floor. The sub-study will occur at Mount Sinai Morningside Cath Lab on the 3rd floor. The study will enroll an estimated total of 70 subjects, 12 of which will also participate in the sub-study. The study is estimated to last 2 years.

DETAILED DESCRIPTION:
All patients will be consented and will undergo Rb-82 rest-stress myocardial perfusion imaging PET with flow quantitation using vasodilator (regadenoson preferred) stressor and cold pressor test and an exercise treadmill test according to standard modified Bruce protocol (if able to exercise).

Only the patients who do not have a recent coronary CT angiography will be consented for undergoing a coronary CT angiography for measurement of plaque burden and quantification of extent and degree of epicardial stenosis.

A small subset of patients who have abnormal flow parameters on PET will be invited to participate in the invasive angiographic validation cohort and will undergo an invasive functional angiography with measurement of FFR, CFR, IMR and Ach-vasoreactivity testing to obtain validation data for PET-guided diagnosis of CMD. A short questionnaire of symptom, suspected diagnosis and planned management will be administered to the treating physician prior to and post-study enrollment.

Patient risk factors, symptoms, health status, medications will be collected using standardized data collection form on study enrollment.

For Aim 2, the cardiac PET findings will be made available to the treating clinician.

A positive PET result for endothelial-independent CMD will be defined as global MBFR <2. A positive PET result for endothelial-dependent CMD will be defined as MBF with cold-pressor test <=40%.

If there was evidence of CMD on cardiac PET, specific treatment recommendations will be made available to the treating physician. These recommendations will include consideration of aspirin, statin and ACE-inhibitors in all patients, beta-blockers (eg: carvedilol 6.25 mg BID with uptitration) as first line, non-dihydropyridine calcium channel blockers (cardizem and verapamil) as second line, and amlodipine (in combination with beta-blocker) or ranolazine as third-line therapy.

Patient symptoms and health status and downstream resource utilization (ER admissions for chest pain, use of other invasive or non-invasive diagnostic procedures for CAD) will be collected at 3 months.

Invasive physiology measurements will be made available to the treating clinician along with recommended management based on INOCA endotype (corMICA trial treatment algorithm) at completion of 3 months.

ELIGIBILITY:
Inclusion criteria:

* Patients with symptoms of exertional angina and/or dyspnea (confirmed on Seattle Angina Questionnaire and Rose Dyspnea Questionnaire)
* Evidence of non-obstructive CAD on CCTA or coronary angiography (no stenosis >50% and/or FFR if performed >0.80)

Exclusion criteria:

* Patients with reduced LVEF (<50%) or diagnosis of cardiomyopathy
* Patients with co-existent moderate or severe valve disease
* Patients with eGFR <30 ml/min/m2
* History of prior coronary revascularization
* Non-coronary indication for CCTA or coronary angiogram determining eligibility
* Contraindications to regadenoson (severe asthma/chronic obstructive pulmonary disease, brady-arrhythmias, or systolic blood pressure <90 mm Hg)
* Inability to provide informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The Seattle Angina Questionnaire (SAQ) | 3 months
  The Seattle Angina Questionnaire (SAQ) is a 7-item self-administered questionnaire with a 4-week recall period measuring health status in patients with CAD across 3 domains: physical limitation (PL), angina frequency (AF), and quality of life (QoL). Full scale from 0-100, with higher score indicating better health outcome.
Rose Dyspnea Scale (RDS) | 3 months
  Rose Dyspnea Scale (RDS) is a 4-item questionnaire with a 1-month recall period that assesses patients' level of dyspnea with common activities. Full scores range from 0 to 4, where 0 indicates no dyspnea with activity and 4 indicates significant limitations due to dyspnea. Higher score indicates poorer health outcomes.
Euro-QOL 5 Dimension Visual Analog Scale (EQ5D-VAS) | 3 months
  Euro-QOL 5 Dimension Visual Analog Scale (EQ5D-VAS) The EQ-5D gives a measure of health-related quality of life. The visual analogue score is a measure of overall self-rated health status with full scale from 0-100. Higher scores indicate better health outcomes.
Number of ER admissions for chest pain per participant | 3 months
  The number of ER admissions for chest pain per participant.
Number of use of other invasive or non-invasive diagnostic procedures for CAD | 3 months
  The number of use of other invasive or non-invasive diagnostic procedures for CAD

SECONDARY OUTCOMES:
The Bruce protocol score | within 3 months of patient enrollment
  Sub group: Treadmill Exercise Stress Test to obtain mean values of exercise capacity (metabolic equivalents, METs) will be assessed for patients with and without CMD as defined on PET.
  The Bruce protocol for exercise test uses a series of calculations to determine a subject's score. This score then indicates physical fitness and the presence of coronary heart disease. The Bruce protocol uses the following calculations: VO2max (ml/kg/min) = 14.76 - (1.379 × T) + (0.451 × T²) - (0.012 × T³) Women: VO2max (ml/kg/min) = 2.94 x T + 3.74 Young Women: VO2max (ml/kg/min) = 4.38 × T - 3.9 Men: VO2max (ml/kg/min) = 2.94 x T + 7.65 Young Men: VO2max (ml/kg/min) = 3.62 x T + 3.91.
Number of participants with METs >=10 METS | within 3 months of patient enrollment
  Prevalence of CMD will be assessed among patients with preserved (METs >=10 METS) and reduced exercise capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Patel, MBBS, MSc, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Morningside, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  For individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link tbd).